CLINICAL TRIAL: NCT06594484
Title: Comparative Analysis of Machine Learning Versus Conventional Models for Predicting Erythrocyte Need in Cardiovascular Surgery
Brief Title: Machine Learning Versus Traditional Scores in Predicting Erythrocyte Need
Status: Completed | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Yuksek, md, Kocaeli City Hospital
Other Study IDs: 2024-6
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Erythrocyte Transfusion; Machine Learning
Keywords: Machine Learning; Cardiovascular Surgery; Perioperative Bleeding; Erythrocyte Transfusion; Predictive Modeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- General Anesthesia Group: The need for ES was recorded in patients undergoing cardiovascular surgery.
  Interventions: Other: Ml Based Algorithm 1; Other: Ml Based Algroithm 2; Other: Bleeding Scores

INTERVENTIONS:
Other: Ml Based Algorithm 1 — The values in the ML algorithm were selected according to logistic regression analysis and the values used in the other six scores tested. The success rate of the constructed networks correct predictions was considered as the success rate of the algorithm. The usefulness of the test was determined through AUROC analysis. Two algorithms were tested in our study. In the first algorithm (ML1), the dependent variable was erythrocyte suspension (ES) consumption, and the independent variables included patients; demographic data, laboratory data, and operational data
Other: Ml Based Algroithm 2 — is an Ml algorithm created by combining commonly used bleeding scores
Other: Bleeding Scores — ACTION CRUSCADE TRACK WILL-BLEED PAPWORTH TRUST ACTAPORT skores used to predict ES need

SUMMARY:
In this study, we compared perioperative bleeding prediction scores with our machine learning-based prediction system in predicting the need for erythrocyte suspension during cardiovascular surgery.

DETAILED DESCRIPTION:
The success of ML algorithms in predicting perioperative blood product use in CABG remains an under-tested topic. Unnecessary preparation of blood products or not being able to supply them when necessary is critical for both patient safety and the effective use of hospital resources [8]. Bleeding amounts and blood product use strategies can vary with institute protocols. Scoring systems that determine the general framework may not perform well due to local factors. ML algorithms can be created locally according to previous patient data of each clinic and can improve themselves with learning mechanisms, suggesting significant potential in this field.

In the current study, a new estimation system created with the ML algorithm was compared with the known estimation systems. Comparing the ML algorithm with 6 different classical scoring systems is important in terms of demonstrating the potential of this technology.

The aim of this study is to investigate whether the model created with ML in predicting perioperative blood product consumption in cardiovascular surgeries is superior to predictive scoring systems that have proven themselves in the literature. Secondary aim is to compare the predictive value of using more than one scoring system in combination.

ELIGIBILITY:
Inclusion Criteria:

* Data from patients who underwent isolated CABG surgeries in the cardiac and vascular surgery operating rooms between 01.01.2023 and 01.01.2024 were evaluated.

Exclusion Criteria:

* Missing Data
* Emergency surgery
* İntraoperative mortality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Complete files from the data of patients undergoing elective cardiac surgery in Kocaeli City Hospital operating rooms will constitute the study data.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
ML algorithm versus traditional scoring in predicting ES needs | During the intraoperative period Cardiac Surgery
  The success of the ML-based algorithm in correctly predicting the ES need will be calculated.

SECONDARY OUTCOMES:
Deterdetermining the most effective method for predicting ES needs using traditional scores | During the intraoperative period Cardiac Surgery
  After comparing the ACTION CRUSCADE TRACK WILL-BLEED PAPWORTH TRUST ACTAPORT scores, the most successful one scoring system will be revealed. The results will be shown numerically with the percentages of predicting the need for ES.

OTHER OUTCOMES:
ML algorithm of combination of scores | During the intraoperative period Cardiac Surgery
  Testing the success of the Ml algorithm based on ACTION CRUSCADE TRACK WILL-BLEED PAPWORTH TRUST ACTAPORT

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmıt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park J, Bonde PN. Machine Learning in Cardiac Surgery: Predicting Mortality and Readmission. ASAIO J. 2022 Dec 1;68(12):1490-1500. doi: 10.1097/MAT.0000000000001696. Epub 2022 May 9. PMID 35544455
- [Background] El-Sherbini AH, Shah A, Cheng R, Elsebaie A, Harby AA, Redfearn D, El-Diasty M. Machine Learning for Predicting Postoperative Atrial Fibrillation After Cardiac Surgery: A Scoping Review of Current Literature. Am J Cardiol. 2023 Dec 15;209:66-75. doi: 10.1016/j.amjcard.2023.09.079. Epub 2023 Oct 21. PMID 37871512
- [Background] Shahian DM, Lippmann RP. Commentary: Machine learning and cardiac surgery risk prediction. J Thorac Cardiovasc Surg. 2022 Jun;163(6):2090-2092. doi: 10.1016/j.jtcvs.2020.08.058. Epub 2020 Aug 24. No abstract available. PMID 32951875
- [Background] Miles TJ, Ghanta RK. Machine learning in cardiac surgery: a narrative review. J Thorac Dis. 2024 Apr 30;16(4):2644-2653. doi: 10.21037/jtd-23-1659. Epub 2024 Apr 24. PMID 38738250
- [Background] Tseng PY, Chen YT, Wang CH, Chiu KM, Peng YS, Hsu SP, Chen KL, Yang CY, Lee OK. Prediction of the development of acute kidney injury following cardiac surgery by machine learning. Crit Care. 2020 Jul 31;24(1):478. doi: 10.1186/s13054-020-03179-9. PMID 32736589